

## **Informed Consent Form**

V3.0 21/09/2019

## The Smoke Free App Smoking Cessation Study

## Name of researchers:

Chief Investigator: Dr Sadia Khan

Co-principal investigators: Dr Pablo Kostelec/Dr Baruah Resham

Additional Investigators: Dr Sofia Cavill, Miss Meera Joshi, Dr Ramyadevi Ravindrane, Dr Ali Kirresh,

Charmaine Bvute, Pranal Gohil

You are consenting to take part of the study, 'Smoke Free app' smoking cessation trial. You may withdraw your participation from this study and your consent at any point, including before and after the study has taken place.

Please initial each box:

IRAS ref: 264547

| I confirm that I have read and understood the patient information sheet (v4.0 21/09/2019) "Smoke Free App Smoking Cessation Study" for this study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. |
|---|
| I confirm that I have had sufficient time to consider whether or not I want to be included in the study. |
| I understand my participation is voluntary and I am free to withdraw at any time, without giving any reason, without prejudice and without my medical care or legal rights being affected. |
| I understand that relevant sections of my medical notes and data collected during the study, may be looked at by individuals from Chelsea and Westminster Hospital NHS Foundation Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. |
| I understand that this consent form will be kept separate from the data and that the researchers will maintain my anonymity throughout the project, including in publication. |
| I agree that the research team notify my general practitioner (GP) of my participation in the Smoke Free App Smoking Cessation Study |
| I agree to take part in the 'Smoke Free app smoking cessation study'. |



| Name of Patient | Date | Signature |
|-------------------------------|------|-----------|
| Name of Person taking consent | Date | Signature |

## Researchers' contact details:

IRAS ref: 264547

Dr Sadia Khan Consultant Cardiologist Chelsea and Westminster Hospital NHS Foundation Trust West Middlesex University Hospital London, TW7 6AF Tel: 0208321 5336

the patient's hospital medical record.

Filling instructions: Please complete one copy for researcher, one for patient and one to be kept in